CLINICAL TRIAL: NCT05664880
Title: A PiLot ClinicaL TrIal of ParicAlcitol for ChroNiC PancrEatitis
Acronym: ALLIANCE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephen Pandol, MD, Director, Basic and Translational Pancreas Research Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00001982; 1R01DK132631-01 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pancreatitis
Keywords: Paricalcitol
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Paricalcitol (Experimental): Participants receive Paricalcitol 2mcg capsule once daily for 12 months.
  Interventions: Drug: Paricalcitol
- Placebo (Placebo Comparator): Participants receive Paricalcitol Placebo capsule matching Paricalcitol once daily for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — 2 MCG Oral Capsule
  Arms: Paricalcitol
Drug: Placebo — Matching capsule to 2 MCG Paricalcitol Oral Capsule
  Arms: Placebo

SUMMARY:
The purpose of this pilot study to examine the feasibility and acceptability of paricalcitol in adults with Chronic Pancreatitis (CP).

DETAILED DESCRIPTION:
Examine the feasibility of a trial to test the effect of paricalcitol through health-related quality of life, imaging, and biomarker analysis in patients with chronic pancreatitis (CP). The study hopes the proposed intervention will improve symptoms based on preclinical evidence that vitamin D analogues have significant and beneficial effects on pancreatitis cancer by blocking certain signaling proteins to reduce pain.

Medical history, concomitant medications, and laboratory test results will be reviewed at all visits by one of the study physicians. In addition, at the beginning and end of the study period, patients will have an MRI to assess condition and DEXA scan to measure bone mineral density, to compare and determine if those receiving paricalcitol have a clinically significant decrease in bone mineral density compared to those receiving placebo for safety. In addition to scans, routine labs will be obtained to assess for any adverse events or safety concerns. Mechanistic specimens for research purposes will be collected at each of the following in person visits: Screening/Randomization, Month 6, Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-75 at time of enrollment
* Diagnosis of Chronic Pancreatitis episode is not attributable to gallstones (i.e. suspected or definite biliary etiology), medications, trauma or autoimmune pancreatitis.
* Ability to take oral medication and be willing to adhere to the dosing regimen
* Normal Calcium levels- 8.5 to 10.2 mg/dL
* Normal Phosphate levels- 2.8 to 4.5 mg/dL
* Normal Parathyroid hormone levels- 10 to 65 pg/mL
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 1 week after the end of Investigational Product administration
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
* No prior pancreatic surgery
* Pancreatic necrosis, if present, is <50% (to be verified by radiologist)
* No involvement in any interventional trials currently or within 6 months of enrollment

Exclusion Criteria:

* Pregnancy or lactation
* History of autoimmune or traumatic pancreatitis, or sentinel attack of acute necrotizing pancreatitis which results in suspected disconnected duct syndrome
* Primary pancreatic tumors - pancreatic ductal adenocarcinoma, suspected cystic neoplasm (>1 cms in size or main duct involvement), neuroendocrine tumors, and other uncommon tumors.
* Pancreatic metastasis from other malignancies
* History of solid organ transplant, HIV/AIDS.
* Abnormal lab values: calcium, phosphate, or parathyroid hormone
* Known isolated pancreatic exocrine insufficiency (e.g. in the absence of any eligible inclusion criteria)
* Participants must not have medical or psychiatric illnesses or ongoing substance abuse that in the investigator's opinion would compromise their ability to tolerate study interventions or participate in longitudinal follow up
* Patients with known abnormal creatinine (GFR < 30) or renal failure (applies to patients with chronic upper abdominal pain of suspected pancreatic origin and suspected CP.
* Known Pregnancy. All participants of childbearing potential, except if post-menopausal [i.e. no menses for ≥2 years] or had a hysterectomy, bilateral tubal ligation/clip (surgical sterilization) or surgical removal of both the ovaries), must have a negative urine or serum B-HCG pregnancy test documented within 2 days prior to any endoscopic or radiologic procedures done for research purposes. Any standard of care tests will follow institutional policies regarding pregnancy test
* Currently incarcerated
* Inability to tolerate MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Examine the feasibility of testing the effect of paricalcitol on health-related quality of life in patients with chronic pancreatitis | End of study (12 Months)
  The proposed trial will examine the feasibility of testing the effect of the vitamin D analogue called paricalcitol (also known as Zemplar), on health-related quality of life, imaging, and biomarkers in patients with chronic pancreatitis (CP).
  Health-related quality of life measurements will be collected via questionnaires to assess overall health, quality of life, and pain. An Acceptability Form will be provided during the last visit to gauge the general acceptability of the intervention.
  Feasibility will be met if ≥75% of enrolled patients complete the 12-month study. There will be a 21-month recruitment period and a one-year treatment period.

SECONDARY OUTCOMES:
Compare the mean change in health related quality of life from baseline across the times points 6 and 12 months between the treatment group and placebo | End of study (12 Months)
  The study will monitor health-related quality of life measures, imaging, and biomarkers to identify potential measures of response to treatment with the intent do develop larger efficacy focused trials.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pandol, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No